CLINICAL TRIAL: NCT00772967
Title: A Double-Blind, Placebo-Controlled, 3-Period Crossover Study to Evaluate the Analgesic Effects of Naproxen and Ultracet in a Walking Model of Osteoarthritis Knee Pain
Brief Title: A Study to Evaluate the Effect of Analgesics on a Walking Model of Knee Pain (0000-105)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-105; 2008_566 (Other: Merck)
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen; Ultracet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo, Naproxen, Ultracet (Experimental): Participants were treated with Placebo for 3 days in Treatment Period 1, Naproxen for 3 days in Treatment Period 2, and Ultracet for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet
- Naproxen, Ultracet, Placebo (Experimental): Participants were treated with Naproxen for 3 days in Treatment Period 1, Ultracet for 3 days in Treatment Period 2, and Placebo for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet
- Ultracet, Placebo, Naproxen (Experimental): Participants were treated with Ultracet for 3 days in Treatment Period 1, Placebo for 3 days in Treatment Period 2, and Naproxen for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet
- Placebo, Ultracet, Naproxen (Experimental): Participants were treated with Placebo for 3 days in Treatment Period 1, Ultracet for 3 days in Treatment Period 2, and Naproxen for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet
- Naproxen, Placebo, Ultracet (Experimental): Participants were treated with Naproxen for 3 days in Treatment Period 1, Placebo for 3 days in Treatment Period 2, and Ultracet for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet
- Ultracet, Naproxen, Placebo (Experimental): Participants were treated with Ultracet for 3 days in Treatment Period 1, Naproxen for 3 days in Treatment Period 2, and Placebo for 3 days in Treatment Period 3. The treatment periods were separated by a 4-6 day break.
  Interventions: Drug: Naproxen; Drug: Placebo; Drug: Ultracet

INTERVENTIONS:
Drug: Naproxen — Naproxen tablets 500 mg twice daily on Day 1, a first dose at t = 0 hrs, and a second dose at t = 12 hrs. Twice daily on Day 2 and 500 mg once daily on Day 3. Walking tests will be performed on Days 1 and 3 of the treatment period.
Drug: Placebo — Placebo capsules twice daily on Day 1, a first dose at t = 0 hrs, and a second dose at t = 12 hrs. Three times daily on Day 2, and 2 capsules on the morning of Day 3. Walking tests will be performed on Days 1 and 3 of the treatment period.
Drug: Ultracet — Ultracet (tramadol/acetaminophen) 37.5/325 mg/mg capsules twice daily on Day 1, a first dose at t = 0 hrs, and a second dose at t = 12 hrs. Three times daily on Day 2, and two 37.5/325 mg capsules on the morning of Day 3. Walking tests will be performed on Days 1 and 3 of the treatment period.

SUMMARY:
This study will evaluate a walking model of osteoarthritis for use in testing of new therapeutic agents. The primary hypothesis is that participants treated with Naproxen or Ultracet will have lower Pain Intensity (PI) than those treated with Placebo during self-paced walks on Day 3 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has osteoarthritis of the knee and primary source of pain is knee
* Females must not be pregnant or nursing and must agree to use birth control throughout the study
* Is willing to limit alcohol and caffeine intake
* Is willing to abstain from smoking during study visits
* Must be able to walk on a treadmill at a pace of at least 1 mile/hour

Exclusion Criteria:

* Has a medical/arthritic disease that would interfere with evaluation
* Is unable to take naproxen or Ultracet
* Has congestive heart failure or angina
* Has a history of stroke
* Has a history of uncontrolled high blood pressure
* Has a history of cancer
* Regularly uses a walker or cane

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Peeva E, Beals CR, Bolognese JA, Kivitz AJ, Taber L, Harman A, Smugar SS, Moskowitz RW. A walking model to assess the onset of analgesia in osteoarthritis knee pain. Osteoarthritis Cartilage. 2010 May;18(5):646-53. doi: 10.1016/j.joca.2009.12.008. Epub 2010 Feb 6. PMID 20175977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 23 June 2008
  Last Patient, Last Visit: 20 November 2008
  2 sites
Pre-assignment Details: Inclusion criteria: Patient has osteoarthritis of the knee and primary source of pain is knee
  Titration schedule for Ultracet® (Acetaminophen 325 mg and tramadol hydrochloride 37.5 mg): twice on Day 1, three times on Day 2, and twice on the morning of Day 3.
  Naproxen tablets 500 mg twice daily on Days 1 and 2 and 500 mg once daily on Day 3.
Groups:
- Placebo, Naproxen, Ultracet: Placebo in Treatment Period 1, Naproxen in Treatment Period 2, Ultracet in Treatment Period 3.
- Naproxen, Ultracet, Placebo: Naproxen in Treatment Period 1, Ultracet in Treatment Period 2, Placebo in Treatment Period 3.
- Ultracet, Placebo, Naproxen: Ultracet in Treatment Period 1, Placebo in Treatment Period 2, Naproxen in Treatment Period 3.
- Placebo, Ultracet, Naproxen: Placebo in Treatment Period 1, Ultracet in Treatment Period 2, Naproxen in Treatment Period 3.
- Naproxen, Placebo, Ultracet: Naproxen in Treatment Period 1, Placebo in Treatment Period 2, Ultracet inTreatment Period 3.
- Ultracet, Naproxen, Placebo: Ultracet in Treatment Period 1, Naproxen in Treatment Period 2, Placebo in Treatment Period 3.
Period: Crossover Treatment 1
Arm/Group | Placebo, Naproxen, Ultracet | Naproxen, Ultracet, Placebo | Ultracet, Placebo, Naproxen | Placebo, Ultracet, Naproxen | Naproxen, Placebo, Ultracet | Ultracet, Naproxen, Placebo
Started | 3 | 5 | 3 | 4 | 4 | 3
Completed | 3 | 5 | 3 | 3 (The withdrawal is not included in any outcomes; but is part of the Adverse Event group for placebo) | 4 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event (Pain) | 0 | 0 | 0 | 1 | 0 | 0
Period: Break 1 (4-7 Days)
Arm/Group | Placebo, Naproxen, Ultracet | Naproxen, Ultracet, Placebo | Ultracet, Placebo, Naproxen | Placebo, Ultracet, Naproxen | Naproxen, Placebo, Ultracet | Ultracet, Naproxen, Placebo
Started | 3 | 5 | 3 | 3 | 4 | 3
Completed | 3 | 4 | 3 | 3 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Crossover Treatment 2
Arm/Group | Placebo, Naproxen, Ultracet | Naproxen, Ultracet, Placebo | Ultracet, Placebo, Naproxen | Placebo, Ultracet, Naproxen | Naproxen, Placebo, Ultracet | Ultracet, Naproxen, Placebo
Started | 3 | 4 | 3 | 3 | 4 | 3
Completed | 3 | 4 | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Break 2 (4-7 Days)
Arm/Group | Placebo, Naproxen, Ultracet | Naproxen, Ultracet, Placebo | Ultracet, Placebo, Naproxen | Placebo, Ultracet, Naproxen | Naproxen, Placebo, Ultracet | Ultracet, Naproxen, Placebo
Started | 3 | 4 | 3 | 3 | 4 | 3
Completed | 3 | 4 | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Treatment 3
Arm/Group | Placebo, Naproxen, Ultracet | Naproxen, Ultracet, Placebo | Ultracet, Placebo, Naproxen | Placebo, Ultracet, Naproxen | Naproxen, Placebo, Ultracet | Ultracet, Naproxen, Placebo
Started | 3 | 4 | 3 | 3 | 4 | 3
Completed | 3 | 4 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (7.92) [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time Weighted Average (TWA) Pain Intensity (PI) on a Numeric Rating Scale (NRS) Due to Self-paced Walks on Day 3
Description: Baseline measurements of participant-specific knee PI were gathered pre-dose on Day 1 from the briskest possible self-pace constant walks on a treadmill over the course of a 20 minute interval. Over this interval PI readings were taken at time points 0,3,6,9,12,15,18 and 20 minutes, rated on an 11-point numeric rating scale (NRS), with 0: No Pain - 10: Worst Pain You Can Imagine. Following a single treatment on Day 3, PI was similarly measured over 20 minute self paced walks at 4 and 6 hrs post-dose. The difference between the TWA (0-20 minutes) PI determined at baseline, and the average of the two TWA (0-20 minutes) PI from the self-paced walks on Day 3 is reported as units on a scale.
Time Frame: Baseline and Day 3
Population: All treated participants who provided baseline and at least one on-treatment observation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo: Participants treated with at least one dose of Placebo
- Naproxen: Participants treated with at least one dose of Naproxen
- Ultracet: Participants treated with at least one dose of Ultracet.
Arm/Group | Placebo | Naproxen | Ultracet
Number analyzed (Participants) | 20 | 21 | 19
units on a scale | -0.927 [-1.52 to -0.33] | -1.54 [-2.12 to -0.96] | -1.73 [-2.34 to -1.12]
Statistical Analysis 1: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p = 0.089, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -0.611, 90% CI [-1.36 to 0.14]
Statistical Analysis 2: Comparison: Placebo vs Ultracet; Test type: Superiority or Other; p = 0.043, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -0.804, 90% CI [-1.57 to -0.04]

2. Secondary Outcome: Change From Baseline in Time Weighted Average (TWA) Pain Intensity (PI) on a Numeric Rating Scale (NRS) Due to Self-paced Walks on Day 1
Description: Baseline measurements of participant-specific knee PI were gathered pre-dose on Day 1 from the briskest possible self-pace constant walks on a treadmill over the course of a 20 minute interval. Over this interval PI readings were taken at time points 0,3,6,9,12,15,18 and 20 minutes, rated on an 11-point numeric rating scale (NRS), with 0: No Pain - 10: Worst Pain You Can Imagine. Following the first treatment on Day 1, PI was similarly measured over 20 minute self-paced walks at 2, 4, and 6 hrs post-dose . The difference between the TWA (0-20 minutes) PI determined at baseline, and the average of the three TWA (0-20 minutes)PI from the self-paced walks on Day 1 is reported as units on a scale.
Time Frame: Baseline and Day 1
Population: All treated participants who provided baseline and at least one on-treatment observation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Naproxen | Ultracet
Number analyzed (Participants) | 21 | 21 | 21
units on a scale | -0.438 [-0.98 to 0.11] | -0.956 [-1.51 to -0.40] | -1.47 [-2.02 to -0.92]
Statistical Analysis 1: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p = 0.048, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -0.518, 90% CI [-1.03 to -0.01]
Statistical Analysis 2: Comparison: Placebo vs Ultracet; Test type: Superiority or Other; p = 0.001, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -1.03, 90% CI [-1.54 to -0.53]

3. Secondary Outcome: Change From Baseline in Time Weighted Average (TWA) Pain Intensity (PI) on a Numeric Rating Scale (NRS) Due to High-paced Walks on Day 1
Description: Baseline measurements of participant-specific knee PI were gathered pre-dose on Day 1 from the briskest possible self-pace constant walks on a treadmill over the course of a 20 minute interval. Over this interval PI readings were taken at time points 0,3,6,9,12,15,18 and 20 minutes,rated on an 11-point numeric rating scale (NRS), with 0: No Pain - 10: Worst Pain You Can Imagine. Following the first treatment on Day 1, PI was similarly measured over a 20 minute high-paced treadmill walk at 5 hrs post-dose. A high-paced walk is the highest pace that can be walked safely for at least 5 minutes that is at a 10-30% higher rate than a self-paced walk. The difference between the TWA (0-20 minutes) PI determined at baseline, and the TWA (0-20 minutes) PI of the high-paced walk on Day 1 is reported as units on a scale.
Time Frame: Baseline and Day 1
Population: All treated participants who provided baseline and at least one on-treatment observation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Naproxen | Ultracet
Number analyzed (Participants) | 21 | 21 | 21
units on a scale | 0.150 [-0.52 to 0.82] | -0.508 [-1.18 to 0.17] | -1.00 [-1.67 to -0.34]
Statistical Analysis 1: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p = 0.052, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -0.658, 90% CI [-1.32 to 0.01]
Statistical Analysis 2: Comparison: Placebo vs Ultracet; Test type: Superiority or Other; p = 0.003, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -1.15, 90% CI [-1.81 to -0.49]

4. Secondary Outcome: Change From Baseline in Time Weighted Average (TWA) Pain Intensity (PI) on a Numeric Rating Scale (NRS) Due to High-paced Walks on Day 3
Description: Baseline measurements of participant-specific knee PI were gathered pre-dose on Day 1 from the briskest possible self-pace constant walks on a treadmill over the course of a 20 minute interval. Over this interval PI readings were taken at time points 0,3,6,9,12,15,18 and 20 minutes, rated on an 11-point numeric rating scale (NRS), with 0: No Pain - 10: Worst Pain You Can Imagine. Following a single treatment on Day 3, PI was similarly measured over a 20 minute high-paced treadmill walk, at 5 hrs post-dose. A high-paced walk is the highest pace that can be walked safely for at least 5 minutes that is at a 10-30% higher rate than a self-paced walk. The difference between the TWA (0-20 minutes) PI determined at baseline, and the TWA (0-20 minutes) PI of the high-paced walk on Day 3 is reported as units on a scale.
Time Frame: Baseline and Day 3
Population: All treated participants who provided baseline and at least one on-treatment observation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Naproxen | Ultracet
Number analyzed (Participants) | 20 | 21 | 19
units on a scale | -0.234 [-0.85 to 0.38] | -1.11 [-1.71 to -0.51] | -1.30 [-1.93 to -0.67]
Statistical Analysis 1: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p = 0.019, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -0.875, 90% CI [-1.56 to -0.19]
Statistical Analysis 2: Comparison: Placebo vs Ultracet; Test type: Superiority or Other; p = 0.007, ANCOVA — 1-sided, alpha = 0.05; Baseline measurement included as covariate: Time-weighted average pain intensity during pretreatment walk; Mean Difference (Final Values) = -1.07, 90% CI [-1.77 to -0.37]

ADVERSE EVENTS:
Time Frame: Adverse experiences (AEs) were collected from the time the consent is signed through the 14 day follow up period after all treatment periods were completed.
Description: AEs were assessed by clinical evaluation including vital signs, physical examination, medical history, clinical laboratory safety assessment (hematology, chemistry, urinalysis), and ECG at timepoints specified in the study. Patients were queried at each visit for any adverse experiences since the previous visit.
Groups:
- Ultracet: Participants treated with at least one dose of Ultracet. Two participants were not treated due to discontinuation.
Arm/Group | Placebo | Naproxen | Ultracet
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Naproxen (N=22) | Ultracet (N=20)
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.